CLINICAL TRIAL: NCT05141279
Title: Contrast Enhanced Mamography in Predicting Response of Breast Cancer Post Neoadjuvant Chemotherapy
Brief Title: Accuracy Of Contrast Enhanced Mamography in Predicting Response of Breast Cancer Post Neoadjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, DMAhmed, Doaa Mahmoud Ahmed, Assiut University
Other Study IDs: CESM in breast cancer
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1: Stable
- 2: Partial response
- 3: Moderate response
- 4: Excellent response
- 5: Complete response

SUMMARY:
The aim of this work to evaluate the accuracy of contrast enhanced spectral mamography in predicting the response to NAC and assessment of residual disease in breast cancer patients

DETAILED DESCRIPTION:
This a prospective series ,will be performed for 50 patients diagnosed by biopsy as breast cancer who will be scheduled for surgery after completing the full coarse of neoadjuvant chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* patient confirmed diagnosed by early breast cancer decided to received neoadjuvant treatment
* locally advanced breast cancer
* operable metastatic breast cancer

Exclusion Criteria:

* patient not candidate for NAC
* contrast allergy
* renal impairment
* pregnancy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 50 patients who will attend to outpatient surgical and oncology clinicS of Assiut university and diagnosed by biopsy as breast cancer
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of contrast enhanced spectral mamography in the predicting of pathological response to NAC and assessment residual disease in breast cancer patients | Basline

SECONDARY OUTCOMES:
Assess best imaging modalities in pedict post neoadjuvant response | Baseline